CLINICAL TRIAL: NCT02065284
Title: Effects of a Home Based Walking Program Using Rhythmic Auditory Stimulation on Walking and Cortical Activation in Patients With Multiple Sclerosis.
Brief Title: Effects of a Home Based Walking Program Using Rhythmic Auditory Stimulation in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: The Kelvin and Eleanor Smith Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HBWP and RAS
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis; Ambulation Difficulty
Keywords: MS; Ambulation
MeSH Terms: conditions — Multiple Sclerosis; Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Walking-Rhythmic Auditory Stimulation (Active Comparator): Walking daily with Rhythmic Auditory Stimulation (RAS) based music for 4 weeks
  Interventions: Other: Rhythmic Auditory Stimulation (RAS)
- Walking- only (Active Comparator): Walking daily with no Rhythmic Auditory Stimulation (RAS) based music for 4 weeks
  Interventions: Other: Rhythmic Auditory Stimulation (RAS)
- Rhythmic Auditory Stimulation (RAS)only (Active Comparator): Listening to based music only daily for 4 weeks
  Interventions: Other: Rhythmic Auditory Stimulation (RAS)

INTERVENTIONS:
Other: Rhythmic Auditory Stimulation (RAS) — Rhythmic Auditory Stimulation (RAS) is a music therapy technique that provides rhythmic auditory cues (like a beat) to help improve patients' movements, especially when walking.
  Other Names: RAS

SUMMARY:
Rhythmic Auditory Stimulation (RAS) is a music therapy technique that provides rhythmic auditory cues (like a beat) to help improve patients' movements, especially when walking.

The purpose of this study is to compare the effect on walking performance of a home based walking program (HBWP) with Rhythmic Auditory Stimulation (RAS), to that of a HBWP without RAS, or to RAS without walking exercise.

A second part of this study will assess the effects of Rhythmic Auditory Stimulation (RAS) on brain activity in patients with Multiple Sclerosis while performing mental imagery of walking.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older
2. diagnosis of MS per Mc Donald criteria
3. Ambulation Index score from 2 to 6 inclusive (clinically observable gait disturbance, whether the subject walks with no, unilateral, or bilateral support)
4. spastic paresis is the main neurologic impairment causing the gait disturbance, per investigator's judgment.

Exclusion Criteria:

1. neurologic impairments other than spastic paresis (e.g. cerebellar ataxia or sensory ataxia), or non-neurologic impairments (e.g. musculoskeletal problems) play a major role in the subject's gait disturbance, per investigator's judgment;
2. treatment for an MS exacerbation in the past 30 days;
3. severe co morbidity precluding participation in the study per investigator's judgment (e.g. severe cardiac or respiratory failure);
4. severe cognitive deficits precluding informed consent or preventing the subject from following study procedures safely
5. contraindication to MRI such as severe claustrophobia and implanted devices such as neurostimulators, pacemakers, aneurysm clips etc.
6. pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Improved gait pattern on gait analysis | 8 weeks
  To compare the effect on gait pattern of a walking program with Rhythmic Auditory Stimulation, to that of a walking program without Rhythmic Auditory Stimulation, or Rhythmic Auditory Stimulation without walking exercise.

SECONDARY OUTCOMES:
Improved walk time on the timed 25 foot walk test | 8 weeks
  To compare the effect on walking performance of a walking program with Rhythmic Auditory Stimulation, to that of a walking program without Rhythmic Auditory Stimulation, or Rhythmic Auditory Stimulation without walking exercise.
Improved distance on the 2 minute walk test | 8 weeks
  To compare the effect on walking performance of a walking program with Rhythmic Auditory Stimulation, to that of a walking program without Rhythmic Auditory Stimulation, or Rhythmic Auditory Stimulation without walking exercise.

OTHER OUTCOMES:
To assess changes in cortical activation induced by Rhythmic Auditory Stimulation in Multiple Sclerosis patients performing mental imagery of walking. | 8 weeks
  Collect functional MRI images while performing guided imagery.

CONTACTS AND LOCATIONS:
Overall Officials: Francois A Bethoux, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Neurological Institute Mellen Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Conklyn D, Stough D, Novak E, Paczak S, Chemali K, Bethoux F. A home-based walking program using rhythmic auditory stimulation improves gait performance in patients with multiple sclerosis: a pilot study. Neurorehabil Neural Repair. 2010 Nov-Dec;24(9):835-42. doi: 10.1177/1545968310372139. Epub 2010 Jul 19. PMID 20643882